CLINICAL TRIAL: NCT05120492
Title: Optimal Management of Extreme Obesity and Severe Knee Osteoarthritis Feasibility Trial
Acronym: OMEOSKO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 41155
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis; Morbid Obesity
Keywords: Arthroplasty, Replacement, Knee; Bariatric Surgery
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity, Morbid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical weight loss (Experimental): sleeve gastrectomy + dietary and lifestyle counseling prior to total knee replacement
  Interventions: Procedure: bariatric surgery followed by total knee replacement
- Standard of Care (No Intervention): dietary and lifestyle counseling prior to total knee replacement

INTERVENTIONS:
Procedure: bariatric surgery followed by total knee replacement — The only intervention is the randomization of the priority of the 2 procedures.
  Arms: Surgical weight loss

SUMMARY:
Does weight loss surgery in patients with morbid obesity prior to knee replacement surgery improve outcomes from knee replacement surgery

DETAILED DESCRIPTION:
RCT involving patients who have severe knee osteoarthritis and have a body-mass index (BMI; the weight in kilograms divided by the square of the height in meters) of 45 to 60 and are randomly assigned to receive dietary and lifestyle counseling for 9 to 13 months followed by total knee replacement (control arm) or sleeve gastrectomy with dietary and lifestyle counseling for 9 to 13 months followed by total knee replacement (treatment arm).

ELIGIBILITY:
Inclusion Criteria:

severe knee osteoarthritis body-mass index of 45 to 60

Exclusion Criteria:

previous total replacement of the same knee, a need for bilateral total knee replacement, and knee pain during the previous week that the patient rated at higher than 60 mm on a 100-mm visual-analogue scale. Also,prior bariatric or complex foregut surgery, significant cardiovascular, pulmonary, renal, liver, gastrointestinal, psychiatric disorders, pregnancy, malignancy within last 5 years, anemia, coagulopathy requiring anti-coagulation therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Pain, mobility and quality of Life | 1 year
  Knee Injury and Osteoarthritis Outcome Score (KOOS4)

SECONDARY OUTCOMES:
EuroQol Group 5-Dimension Self Report Questionnaire (EQ-5D) | 1 year
  assessing quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada